CLINICAL TRIAL: NCT03663088
Title: Pilot Study for a Randomized Controlled Clinical Trial on the Effect of Global Postural Re-education in the Treatment of Idiopathic Scoliosis: a Feasibility Study
Brief Title: Effect of Global Postural Re-education in Idiopathic Scoliosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the COVID-19 pandemic
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Carole Fortin, Professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StJustineH_CFortin
Record Dates: First submitted 2018-08-02; First posted 2018-09-10 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Scoliosis
Keywords: Physiotherapy; Global postural re-education; Cobb angle; Posture; Back pain; Participation
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPR-A (Active Comparator): The 6-months supervised GPR-A group will receive a 1-hour-long individual session once a week plus a home program (1 or 2 exercises, 2 times a week).
  Interventions: Other: GPR-A
- GPR-B (Experimental): The 6-months supervised GPR-B group will receive a 1-hour long individual session once per two weeks alternately with a 1-hour-long class of exercises once per two weeks plus a home program (1 or 2 exercises, 2 times a week).
  Interventions: Other: GPR-B

INTERVENTIONS:
Other: GPR-A — Standard Global postural re-education physiotherapy scoliosis specific exercises
  Arms: GPR-A
Other: GPR-B — Experimental Global postural re-education physiotherapy scoliosis specific exercises combining individual and class exercises
  Arms: GPR-B

SUMMARY:
In North America, children and adolescents with idiopathic scoliosis (IS) are rarely referred for a rehabilitation program whereas the European guidelines stated that scientific evidences concerning scoliosis specific physiotherapy exercises were strong enough to recommend the use of these exercises at an early stage. The objectives of this pilot study is to assess feasibility of conducting a larger randomized control trial (RCT) on the effect of global postural re-education (GPR) on scoliosis progression (Cobb angle) and posture, back pain and participation and to assess the equivalence of two groups of GPR interventions. A convenience sample of 60 adolescents with IS (Cobb angle 15º-50º, Risser sign ≤3) will be recruited at CHU Sainte-Justine. Participants will be randomly allocated to GPR-A (individual sessions once a week) or GPR-B (individual sessions once per two weeks alternately with class exercises once per two weeks) for 6 months. After 6 months, groups will be interchanged for another 6 months. Feasibility outcomes will be recruitment rate, consent rate, completion rate and adherence to treatment at 12 months. The primary outcome of the effect of GPR will be the Cobb angle. Secondary outcomes will be: posture, back pain and participation at 6 and 12 months. Statistical analyses: For feasibility, percentage of eligible patients recruited, percentage of recruited patients who completed the trial and adherence to treatment will be calculated. For the preliminary effects of GPR, linear mixed-models will be used to assess differences in groups' changes from baseline, to 6 and 12-month while adjusting for covariates (age, Risser, adherence). Separate analyses will be conducted for each outcome.

ELIGIBILITY:
Inclusion Criteria:

* aged between 8 and 16 years old,
* Cobb angle between 15º and 50º,
* a Risser sign ≤3 (skeletal growth incomplete),
* having recent x-rays (4-6 weeks),
* ability to travel weekly to attend GPR interventions

Exclusion Criteria:

* patients who are planning surgery or have had surgery,
* previous regular physiotherapy or other conservative treatment (chiro, osteopathy),
* worn a brace for at least three months prior to GPR interventions,
* scheduled for clinic follow-up later than in 6±2 months,
* or to be discharged before 12 months.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Cobb angle | 6 and 12 months
  Change in the frontal radiologic measure of scoliosis: a decrease in Cobb angle by more than 5 degrees indicate improvement

SECONDARY OUTCOMES:
Posture: shoulder elevation | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The angle formed between a line drawn between the left and right coracoid process markers, and the horizontal: a decrease of this angle indicate improvement
Posture: right waist angle | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The angle formed by lines drawn from the upper end of the waist to the center of the waist, and from the cent Clinical Photographic Postural Assessment Tool: The angle formed by lines drawn from the upper end of the waist to the center of the waist, and from the center of the waist to the lower end of the waist on the right side: more symmetry with the left side indicate improvement
Posture: left waist angle | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The angle formed by lines drawn from the upper end of the waist to the center of the waist, and from the cent Clinical Photographic Postural Assessment Tool: The angle formed by lines drawn from the upper end of the waist to the center of the waist, and from the center of the waist to the lower end of the waist on the left side: more symmetry with the right side indicate improvement
Posture: thoracic scoliosis | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The angle formed by lines drawn from the upper end-vertebra to the apex of the thoracic scoliosis curve and from the apex to the lower end-vertebra of the curve: decrease of this angle indicate improvement
Posture: lumbar scoliosis | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The angle formed by lines drawn from the upper end-vertebra to the apex of the thoracolumbar or lumbar scoliosis curve, and from the apex to the lower end-vertebra of the curve: decrease of this angle indicate improvement
Posture: frontal trunk list | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The horizontal distance between C7 and a vertical line drawn from S1: decrease of this measure in millimeter indicate improvement
Posture: frontal pelvic tilt | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The angle formed between the line joining the two anterior superior iliac spine (ASIS) and the horizontal: decrease of this angle indicate improvement
Posture: right sagittal pelvic tilt | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The angle formed between the horizontal and the line joining the posterior superior iliac spine (PSIS) and ASIS on the right side: an angle between 20 and 30 degrees indicate a normal value and a better symmetry between right and left side indicate improvement
Posture: left sagittal pelvic tilt | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The angle formed between the horizontal and the line joining the PSIS and ASIS on the left side: an angle between 20 and 30 degrees indicate a normal value and a better symmetry between right and left side indicate improvement
Posture: scapula asymmetry | 6 and 12 months
  Clinical Photographic Postural Assessment Tool: The angle formed by a line drawn from the left and right inferior angles of the scapula and the horizontal: decrease of this angle indicate improvement
Change in back pain | 6 and 12 months
  Change in the intensity (score) of back pain on the Numeric Pain Rating Scale score (0 no pain to 10 very important pain), lower value indicate improvement.
Change in score of The youth version of the Child & Adolescent Scale of Participation | 12 months
  Change in score of The youth version of the Child & Adolescent Scale of Participation (CASP): The CASP questionnaire has 20 items x 4 levels from 1 (unable to participate) to 4 (age expected/full participation) with a maximum of 80 points. Higher value indicate improvement (better participation).

OTHER OUTCOMES:
Recruitment rate | 12 months
  Percentage of eligible patients recruited: 70% of participants recruited indicate good recruitment rate
Completion rate | 12 months
  Percentage of recruited participants who completed the trial: 75% of completion indicate good completion rate
Adherence (compliance) with GPR treatment in terms of collaboration, presence and implication in home exercises | 12 months
  Adherence with GPR treatment will be measured by the physiotherapists using the validated 3-item Sport Injury Rehabilitation Adherence Scale (SIRAS, were total score varies from 3 (low adherence) to 15 (high adherence)). We will also compute presence/absence to therapy and we will use a patient/parent logbook for home exercises. Good adherence (compliance) to treatment will be achieved if a participant has a score of at least 12 out of 15 on the SIRAS 80 % of the treatment sessions, is present to therapy 80% of the sessions and completes home exercises 80% of the time.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Fortin, Ph.D., Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided